CLINICAL TRIAL: NCT07297407
Title: PREVENTION-IN-PD - Development of a Multidomain Lifestyle Intervention Study for Prodromal and Clinical Parkinson's Disease
Brief Title: Prevention-in-PD-Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: University Hospital, Bonn (Other); University of Cologne (Other); Philipps University Marburg (Other); University of Kiel (Other)
Responsible Party: Principal Investigator, Eva Schaeffer, PD Dr. Eva Schäffer, University Hospital Schleswig-Holstein
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: D538-25
Record Dates: First submitted 2025-09-16; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Parkinson's Disease (PD)
Keywords: lifestyle; exercise; nutrition; cognitive training; sleep
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multidomain lifestyle intervention (Experimental): Multidomain lifestyle intervention including physical and cognitive training, sleep and nutrition counceling
  Interventions: Other: Multidomain lifestyle intervention

INTERVENTIONS:
Other: Multidomain lifestyle intervention — Lifestyle intervention including physical and cognitive training, nutritional and sleep counseling

SUMMARY:
The goal of this clinical trial (feasibility study) is to learn if a multimodal lifestyle program can improve adherence to recommended lifestyle changes in people with REM Sleep Behavior Disroder (RBD) or Parkinson's disease (PD).

The main question it aims to answer is if individuals with RBD oder PD can follow a combined lifestyle program over six months Participants will take part in a six-month intervention program that includes: Physical training, Mediterranean diet counseling, Sleep counseling and cognitive training.

The program will be supported by psychoeducation, skills training, and personalization to make it practical and motivating.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is becoming more common worldwide, but there are still no treatments that can slow down or stop the disease. Lifestyle changes such as more physical activity, a healthy diet, good sleep, and mental training may help slow down the progression of the disease. However, it is often difficult for people to follow several lifestyle changes at the same time, and no study has yet tested how well this works in Parkinson's.

The PREVENTION-IN-PD study will test a new lifestyle program for people with PD and people with REM Sleep Behavior Disorder (RBD, at risk for developing Parkinson's Disease) in Germany. Over six months, participants will receive support in four areas: exercise, Mediterranean diet, sleep habits, and cognitive training. The program is designed to be practical, personalized, and motivating.

The main goal is to see whether people with PD and RBD can stick to these lifestyle changes over time. The study will also look at potential early effects on symptoms, quality of life, and overall health. If successful, this project will be the first step toward making lifestyle programs an important part of Parkinson's care in Germany and beyond.

ELIGIBILITY:
Inclusion Criteria:

* All participants: ability to perform informed consent; age 30-85
* RBD group: polysomnographic proven diagnosis of isolated REM sleep behavior disorder (iRBD)
* PD group: early to moderate disease (Hoehn & Yahr stage 1-2.5), diagnosis according to the Movement Disorder Society diagnostic criteria for clinical Parkinson's Disease
* Agreement to participate in group sessions and online meetings

Exclusion Criteria:

* dementia (Mini Mental Score, MMSE < 19 points) (MMSE is specifically chosen here to avoid too frequent repetitions of the MoCA, which is used as an outcome parameter for the interventional trial)
* physical inability to perform exercise training or other trainings as judged by a physician
* manifest (severe) depression (Beck Depression Inventory, BDI-II > 29 points)
* participation in other interventional trials
* other significant diseases of the central nervous system
* Planned change in medication within the following 6 months

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Adherence | From enrollement to the end of the intervention after 6 months.
  Adherence to the multimodal lifestyle intervention program is objectively recorded as the primary outcome parameter (participation in the planned training sessions in %). In addition, subjective adherence is recorded (assessment of the implementation of lifestyle measures in everyday life using a Likert scale).

IPD SHARING:
Plan to Share IPD: Undecided